CLINICAL TRIAL: NCT03662295
Title: Stroke-like Migraine Attacks After Radiation Treatment (SMART) Syndrome Language Intervention
Status: Completed | Type: Observational
Sponsor: Quality Living, Inc. (Other)
Responsible Party: Principal Investigator, Karen Hux, Director of Research, Quality Living, Inc.
Other Study IDs: SMART
Record Dates: First submitted 2018-09-03; First posted 2018-09-07 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Migraine Disorders; Aphasia
Keywords: Cognitive Impairment
MeSH Terms: conditions — Migraine Disorders; Aphasia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Language treatment — Individual speech-language therapy sessions totaling 1.5 to 2.5 hours five days per week. Intervention activities include performing oral and written confrontation and responsive naming, writing single words to dictation, reading single words and sentences aloud, and generating written and spoken picture descriptions.

SUMMARY:
Stroke-like migraine attacks after radiation therapy-also known as SMART syndrome-constitute a rare condition typically characterized by headache, seizures, vision abnormalities, hemiparesis, and aphasia. The condition usually resolves within a few days or weeks of onset with no residual impairments. However, resolution in some cases extends over a period of months rather than weeks and may be incomplete. The purpose of this case report is to provide an in-depth description of the progression of changes in cognitive and language functioning for a person exhibiting SMART syndrome characterized by slow recovery.

ELIGIBILITY:
Inclusion Criteria:

* exhibit cognitive and language deficits secondary to SMART syndrome
* be a former or current client of Quality Living, Inc., Omaha, Nebraska
* be a native speaker of English

Exclusion Criteria:

-

Ages: 19 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: One adult with SMART syndrome will participate in this study. The person will have cognitive and language deficits typical of those exhibited by people with SMART syndrome. Given the rarity of the disorder, only one participant is anticipated.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Standardized assessment | Change from baseline at 6 months
  Aphasia Quotient of the Western Aphasia Battery - Revised

SECONDARY OUTCOMES:
Spoken picture description | Change from baseline at 6 weeks, 10 weeks, 14 weeks, 20 weeks, and 26 weeks
  Spoken language sample elicited through a request to describe events depicted in a Norman Rockwell drawing.
Written picture description | Change from baseline at 6 weeks, 10 weeks, 14 weeks, 20 weeks, and 26 weeks
  Written language sample elicited through a request to write about events depicted in a Norman Rockwell drawing.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hux, Ph.D., Principal Investigator — Quality Living, Inc., Omaha, Nebraska
Locations (1):
- Quality Living, Inc., Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No